CLINICAL TRIAL: NCT03974854
Title: Evaluation of Polychemotherapy With XELOXIRI-3 in Elderly or Frail Patients With Advanced Pancreatic Adenocarcinoma (ALIX)
Brief Title: Evaluation of Polychemotherapy With XELOXIRI-3 in Elderly or Frail Patients With Advanced Pancreatic Adenocarcinoma
Acronym: ALIX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2018/395
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Irinotecan; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: XELOXIRI-3 (Experimental): capecitabine 625 mg/m2 twice daily on days 1-7 oxaliplatine 85 mg/m2 on Day 1 irinotecan 90 mg/m2 on Day 3, every 14 days
  Interventions: Drug: XELOXIRI-3
- Arm B: Gemcitabine (Active Comparator): 1000 mg / m2 on D1, D8 and D15, every 28 days
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: XELOXIRI-3 — chemotherapy with XELOXIRI-3 regimen
  Other Names: Capecitabine; Oxaliplatine; Irinotecan
  Arms: Arm A: XELOXIRI-3
Drug: Gemcitabine — chemotherapy with Gemcitabine regimen
  Arms: Arm B: Gemcitabine

SUMMARY:
Current standard of care for patients with metastatic Pancreatic Ductal AdenoCarcinoma (PDAC) is chemotherapy, preferential regimen being FOLFIRINOX (5-fluorouracil, leucovorin, irinotecan, and oxaliplatin). Due to more hematologic (neutropenia) and gastrointestinal toxicities, FOLFIRINOX is only administered in fit patients (age < 75 years, ECOG Performance status 0-1, and bilirubin < 1.5 ULN).

However, elderly or frail patients represent more than half of patients with PDAC and are treated with gemcitabine monochemotherapy. Maintaining more than one drug (polychemotherapy) may improve survival and quality of life in this population.

ALIX is a non-comparative randomized 2:1 phase II study. This study will assess the efficacy and safety of the polychemotherapy with XELOXIRI-3 versus gemcitabine as first-line chemotherapy in elderly or frail patients with locally advanced or metastatic PDAC.

ELIGIBILITY:
Main Inclusion Criteria :

* Histologically proven pancreatic ductal adenocarcinoma
* Locally Advanced or metastatic disease
* Measurable disease according to RECIST v1.1 criteria
* Age ≥ 75 years;

OR age between 65 and 75 years AND with at least one frailty contraindication to the administration of chemotherapy with FOLFIRINOX:

* Eastern Cooperative Oncology Group Performance status (ECOG-PS) 2
* Total serum bilirubin > 1.5 ULN (biliary drainage allowed)
* Clinico-biological frailty criteria:
* weight loss > 10% in 6 months or > 5% in 1 month
* or body mass index (BMI) ≤ 21
* or serum albumin < 30 g/L
* or ADL (Activities of Daily Living) score < 6

  * Eligible for gemcitabine as first-line chemotherapy
  * Registration in a national health care system
  * Written informed consent obtained from the patient prior to performing any protocol-related procedures

Main Exclusion Criteria:

* Age < 65 years
* Localized non-metastatic cancer
* ECOG-PS 3-4
* Previous treatment For advanced stage (locally advanced or metastatic): chemotherapy, radiochemotherapy; For localized stage: FOLFIRINOX chemotherapy (neoadjuvant or adjuvant); adjuvant chemotherapy with gemcitabine before relapse is permitted (provide it has been administered more than 6 months before)
* Uncontrolled intercurrent cardiovascular disease
* Known or suspected allergy or hypersensitivity to any of the study drugs (capecitabine, oxaliplatin, irinotecan, gemcitabine)
* Bowel obstruction or sub-obstruction or impossible oral treatment
* Prior peripheral neuropathy of grade ≥ 2
* Known complete dihydropyrimidine dehydrogenase (DPD) or UDP-glycosyltransferase 1 polypeptide A1 (UGT1A1) deficiency
* Inadequate hematological, hepatic, and renal functions
* Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs (Adverse Events) or compromise the ability of the patient to give written informed consent
* Tutelage or guardianship
* Diagnosis of any second malignancy within the last 2 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri
* Current participation in another clinical trial using therapeutic experimental agents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
6 months Progression-Free Survival (PFS) rate | 6 months after the date of initiation of treatment (1st day of 1st cycle of chemotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Angélique VIENOT, Dr, Principal Investigator — University Hospital of Besançon
Locations (5):
- France (5):
  - University Hospital of Besançon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard
  - CH Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - CHU Reims, Reims

IPD SHARING:
Plan to Share IPD: No